CLINICAL TRIAL: NCT06345495
Title: High Dose Ruxolitinib and Allogeneic Stem Cell Transplantation in Myelofibrosis Patients With Splenomegaly
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0899; NCI-2024-02814 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Splenomegaly; Myelofibrosis
MeSH Terms: conditions — Splenomegaly; Primary Myelofibrosis | interventions — ruxolitinib; Levetiracetam; eltrombopag; Busulfan; romiplostim; fludarabine phosphate; fludarabine; Cyclophosphamide; Mesna; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib and Allogeneic Stem Cell Transplantation (Experimental): Participants will be asked to receive study drugs and a stem cell transplant and attend study visits, at which various tests and procedures will be performed. Participants are expected to receive treatment for about 100 days, followed by a year of follow-up.
  Interventions: Drug: Ruxolitinib; Procedure: Allogeneic Stem Cell Transplantation; Drug: Levetiracetam; Drug: Eltrombopag; Drug: Busulfan; Drug: Romiplostim; Drug: Fludarabine phosphate; Drug: Cyclophosphamide; Drug: Mesna; Drug: Tacrolimus

INTERVENTIONS:
Drug: Ruxolitinib — Given by PO
  Other Names: Jakafi; INCB018424; INC424
Procedure: Allogeneic Stem Cell Transplantation — Given by Transplant
  Other Names: Autologous stem cell transplant; Cord Blood
Drug: Levetiracetam — Given by PO
Drug: Eltrombopag — Given by PO
  Other Names: Promacta®
Drug: Busulfan — Given by IV
  Other Names: Busulfex™; Myleran®
Drug: Romiplostim — Given by IV
  Other Names: AMG 531; Nplate
Drug: Fludarabine phosphate — Given by IV
  Other Names: Fludarabine; Fludara®
Drug: Cyclophosphamide — Given by IV
  Other Names: Cytoxan®; Neosar®
Drug: Mesna — Given by IV
  Other Names: Mesnex™
Drug: Tacrolimus — Given by IV or PO
  Other Names: Prograf®

SUMMARY:
To learn if giving ruxolitinib and busulfan before a stem cell transplant can help to reduce spleen size and help the transplant to succeed.

DETAILED DESCRIPTION:
Primary Objective

1) Compare the proportion of patients alive, disease free, engrafted, and without poor graft function at 100 days post-transplant with the historical rate of 45%.

Secondary Objectives:

1. Overall survival
2. Progression-free survival
3. Graft vs host disease relapse free survival
4. Relapse rate
5. Non-relapse Mortality
6. Time to Neutrophil and platelet engraftment
7. Time to red cell transfusion independence
8. Graft failure
9. Acute and chronic GVHD
10. Grade 3 -5 Toxicity
11. Incidence of poor graft function5
12. Need for growth factors (myeloid or thrombopoietic) at 100 days
13. Spleen response around day -7, -1, 30, and 100 days
14. Need for transfusions at 100 days
15. Time to discontinuation of immunosuppressives

Exploratory Objectives:

1. Immune reconstitution
2. Cytokine profile

ELIGIBILITY:
Inclusion Criteria:

1. Participants 18 years to less than or equal to 75 years.
2. Able to provide written consent.
3. Primary or secondary Myelofibrosis (may have received Jak inhibitors including ruxolitinib)
4. Enlarged spleen by palpation or imaging. For the purpose of this study, splenomegaly is defined as any clinically palpable spleen or spleen larger than 12 cms on imaging.
5. Has a fully matched (8/8:HLA A, B, C, DRB1) related or matched unrelated donor.
6. Adequate renal function, including:

   a. Serum creatinine </= 1.5 mg/dL or estimated Glomerular Filtration Rate (eGFR using the CKI-EPI equation) >/= 40 ml/min/1.73 m2.
7. Adequate liver function, including:

   1. ALT/AST </= 3 x ULN
   2. Direct bilirubin </= 1mg/dL
   3. No history of liver cirrhosis. No ascites.
8. Female participants of childbearing potential must have negative results for a serum pregnancy test. Female participants must agree to not breastfeed during the study and for 3 months post-completion of the study therapy.
9. Subjects who are of childbearing potential, sexually active, and at risk of pregnancy must agree to use a highly effective method of contraception for the duration of the active treatment and at least 3 months post-completion of the study therapy. Highly effective methods of contraception include the following:

   1. Hormonal contraception (i.e., birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
   2. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of study agent administration. Men who are able to have children must use effective birth control while on the study. If the male participant fathers a child or suspects that he has fathered a child while on the study, he must immediately notify his doctor.

Exclusion Criteria:

1. Positive beta HCG in females of child-bearing potential defined as not postmenopausal for 24 months or no previous surgical sterilization or lactating females.
2. Ejection fraction <40%
3. Corrected DLCO < 50%
4. Evidence of other clinically significant uncontrolled condition(s) including, but not limited to:

   1. Uncontrolled and/or active systemic infection (viral, bacterial or fungal)
   2. Active hepatitis B virus (HBV), hepatitis C (HCV), HIV or TB infection or requiring treatment for the same.
   3. Thrombosis including MI, Stroke, PE, DVT in the past 6 months

Note: subjects with serologic evidence of prior vaccination to HBV (i.e. hepatitis B surface (HBs) antigen negative-, anti-HBs antibody positive and anti-hepatitis B core (HBc) antibody negative) or positive anti-HBc antibody from intravenous immunoglobulins (IVIG) may participate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Uday Popat, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org